CLINICAL TRIAL: NCT02146950
Title: European Active Surveillance Study of LCS12
Acronym: EURAS_LCS12
Status: Active, not recruiting | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: ZEG2013_10; 16470 (Other: Bayer AG); EUPAS6476 (Registry Identifier: EUPAS Register)
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Contraception
Keywords: LCS-12; Intrauterine Device (IUD); Intrauterine System (IUS); Levonorgestrel; Pearl Index; Hormonal Contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- LCS12: New users of LCS12
- Mirena: New users of Mirena
- Copper IUD: New users of copper IUDs
- Kyleena: New users of Kyleena
- Other hormonal IUD (OHIUD): New users of other hormonal IUDs (e.g. Levosert, Fibroplant)

SUMMARY:
This study is designed to investigate whether LCS12 is associated with an increased risk of unintended pregnancy compared to Mirena and to copper IUDs. The objective is to assess among new users the risks of certain events (e.g. contraceptive failure rate, ectopic pregnancy, uterine perforation, and PID) associated with the use of LCS12 compared with the established hormonal IUD Mirena, and compared with established copper IUDs during standard clinical practice. In addition, drug utilization patterns will be described.

DETAILED DESCRIPTION:
Intrauterine contraceptive methods, such as Mirena and copper IUDs, have a high contraceptive efficacy. LCS12 is a new intrauterine system which, like Mirena, contains levonorgestrel (LNG), but the T-body dimensions and insertion tube diameter of LCS12 are smaller.

Because there is a lack of comparative data between LCS12 and other intrauterine contraceptives, it is unclear whether there are differences in contraceptive failure rates between LCS12 and either Mirena or copper IUDs. In addition, any transcervical procedure, including the insertion of an intrauterine device, is potentially associated with the risk of infection/inflammation.

EURAS-LCS12 is a prospective, controlled, non-interventional, active surveillance cohort study with three user cohorts: LCS12, Mirena and copper IUDs. Study participants will be recruited by a network of health care professionals and will be followed up through active surveillance to collect information regarding the outcomes of interest and major safety outcomes.

All self-reported clinical outcomes of interest will be validated by health care professionals. The primary endpoint is unintended pregnancy. Secondary endpoints are ectopic pregnancy, uterine perforation, and pelvic inflammatory disease (PID).

Study Amendment (Approved by PRAC on September 29, 2016):

The primary objective of the study is to assess the contraceptive failure risk of Jaydess, Mirena, and copper IUD use in a study population that is representative of the real users of the individual IUDs. Interim analysis showed a high proportion of IUD users in the age group >= 40 years of age. Given the fact that the age distribution remains considerably skewed, and that the Pearl Index is influenced by the age of participants, the independent Safety Monitoring and Advisory Council decided to suggest to narrow the study inclusion criteria, i.e. an age restriction to <40 years old at study entry was suggested for the remaining recruitment phase.

All analyses regarding unintended pregnancies (including ectopic pregnancies) will be conducted using the complete cohorts (i.e. including study participants aged 40 years and older). In addition, these analyses will be done including only women in the age group below 40 years. Further age-stratified analyses of these outcomes are also planned.

Study Amendment (Approved by PRAC in February, 2018):

In addition, due to concerns regarding the influence of the use of hormonal IUDs on neuropsychiatric disorders, the PRAC requested to investigate the baseline risk as well as the risk under exposure of IUDs within the EURAS-LCS12 study.

The baseline questionnaire will capture information on the history of anxiety, panic attacks, mood swings/depression, persistant difficulties with sleeping and restlessness (further on referred to as "neuropsychiatric complaints") for all newly recruited users after ethical approval of the revised questionnaire. Neuropsychiatric complaints that occur under exposure to an IUD reported by the study participant during the follow-up will be validated with the treating physician, if applicable, in the same manner as other outcomes of interest.

Furthermore, the study will be also conducted in Spain and Italy to be able to fulfil study goal in time, as the recruitment of Jaydess users is lower than expected due to the recent launch of another hormonal IUS (Kyleena) which is licensed for contraception for 5 years.

Study amendment (Approved by PRAC in October 2019):

In the course of the study, another hormonal IUD ( 'Kyleena') was launched in 2017 which has the same dimensions as LCS12, but a higher LNG content, and is approved for use up to 5 years. The initial LNG release rates are approximately 14 µg/24h for LCS12, 20 µg/24h for Mirena and 17.5 µg/24h for Kyleena. New users of Kyleena were continuously enrolled in the study since the market introduction and are categorized as 'other hormonal IUD'. However, with increasing usage of Kyleena and enrolment into the EURAS-LCS12 study, the Safety Monitoring and Advisory Council endorsed inclusion of Kyleena as an official cohort to the study to better understand current routine clinical practice. As comparative data on contraceptive failure between Kyleena and Mirena based on routine clinical practice are not available at present, the comparison of contraceptive failure rates between Kyleena and Mirena / copper IUDs was added as an additional secondary outcome to the EURAS-LCS12 study.

As the liscensed duration of use for Kyleena is 6 years, two additional follow-up questionnaires will be sent to eligible users of Kyleena, Mirena and copper IUDs to assess the complete life-cylce of the products.

Study amendment (Approved by PRAC in February 2022):

The purposes of this amendment no. 5 include an adaption of the timelines and recruitment target to allow for completion of the recruitment for the LCS12 cohort, and a merge of the final study report I (including LCS12 3-year results) and II (including Kyleena 5-year results). Further, the statistical methods used for confounder assessments will be adapted to address the imbalances between the cohorts. Finally, the inclusion of copper IUDs will be limited to 30% of current recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Women aged below 40 years who have a new IUD inserted (LCS12, Kyleena, Mirena, copper IUD, or any other hormonal IUD)
* Women who are willing to participate in the active surveillance

Exclusion Criteria:

* Women aged 40 or older at insertion day
* Women who are currently enrolled in an interventional trial on IUD use can not participate

Max Age: 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Only women are eligible for enrolment
Study Population: Women using an intrauterine system/device (hormonal IUS or copper IUD)
Sampling Method: Non-Probability Sample
Enrollment: 97265 (Actual)
Dates: Start 2014-06-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Contraceptive failure (LCS12 vs. Mirena and copper IUDs) | within 3 years

SECONDARY OUTCOMES:
Pelvic inflammatory disease (PID) | within 3 - 5 years
Ectopic pregnancy | within 3 - 5 years
Uterine perforations | within 3 - 5 years
Contraceptive failure (Kyleena vs. Mirena and copper IUDs) | within 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Klaas Heinemann, PhD, MD, MSc, MBA, Principal Investigator — Center for Epidemiology and Health Research Berlin
Locations (1):
- Center for Epidemiology and Health Research Berlin, Berlin, Germany

REFERENCES:
- [Result] Boehnke T, Eggebrecht L, Viet M, Heinemann K, Bauerfeind A. How did regional lockdowns during the COVID-19 pandemic affect recruitment into a large multinational cohort study of intrauterine device users? Contraception. 2023 Jul;123:110003. doi: 10.1016/j.contraception.2023.110003. Epub 2023 Mar 12. PMID 36918064
- [Result] Eggebrecht L, Bauerfeind A, Boehnke T, Rizzo M, Hagemann C, Lange J, Viet M, Pauls K, von Stockum S, Klinghardt M, Heinemann K. Population characteristics of intrauterine device users in real-world clinical practice across Europe - insights from the EURAS-LCS12 study. Contracept Reprod Med. 2025 Mar 14;10(1):20. doi: 10.1186/s40834-025-00353-8. PMID 40087799
- [Result] Boehnke T, Bauerfeind A, Eggebrecht L, Cellier C, Lange JA, Heinemann K, Madden T. Does the shape of the copper intrauterine device play a role in expulsion? Results from the ongoing European Active Surveillance Study on LCS12. Contraception. 2024 Dec;140:110444. doi: 10.1016/j.contraception.2024.110444. Epub 2024 Mar 27. PMID 38552821
- See also: Boehnke T, Bauerfeind A, Hagemann C, Lange JA, Heinemann K, Intrauterine device prescribing patterns and types in Europe - a cross-sectional analysis of the European Active Surveillance LCS12 Study. European Gynecology & Obstetrics — https://www.egojournal.eu/wp-content/uploads/journal/2022/4.1/29/29-40.pdf